CLINICAL TRIAL: NCT03499626
Title: Phase 1b Open Label Dose Assessment Study of ASLAN001 (Varlitinib) in Patients With Advanced/ Metastatic Hepatocellular Carcinoma (HCC) With an Expansion Cohort in HCC Patients Expressing HER3 Who Have Progressed on First Line Sorafenib or Lenvatinib
Brief Title: Phase 1b of ASLAN001 (Varlitinib) in Patients With Advanced/ Metastatic Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/01227; HC01/12/16 (Other: NUH)
Record Dates: First submitted 2018-04-08; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Advanced/ Metastatic Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASLAN001 (Experimental): A 3+3 study de-escalating dose design will be employed for dose determination. Subjects will receive treatment in 21-day cycles until disease progression, intolerable toxicities or withdrawal of consent.
  Interventions: Drug: ASLAN001

INTERVENTIONS:
Drug: ASLAN001 — Starting dose at 300mg BD Dose level +1: 400mg BD (which is the target dose for this study)
  Dose reduction of ASLAN001 in event of adverse events grade 2 and above:
  Dose level -1: 200mg BD Dose level -2: 100mg BD
  Other Names: Varlitinib

SUMMARY:
This is a single-arm, allocation open label study. Phase 1 is a dose-finding phase in patients with advanced/ metastatic hepatocellular carcinoma (HCC) who have progressed on first line Sorafenib or Lenvatinib.

The primary objective of this study will be to establish the maximal tolerable dose (MTD) of ASLAN001 (Varlitinib) in the study population

The secondary objectives include:

1. To evaluate the efficacy of ASLAN001 (Varlitinib), as measured by duration of response (DoR), progression free survival (PFS), overall survival (OS) and disease control rate (DCR)
2. To assess the ORR, DoR, PFS, DCR and OS by tumor EGFR/HER2/HER3/HER4 status
3. To identify tumor and host biomarkers predictive of treatment response or toxicity to ASLAN001.

DETAILED DESCRIPTION:
* There are currently no effective and approved second line treatment options for advanced/ metastatic HCC.
* ASLAN001 (Varlitinib) is a small molecule tyrosine kinase inhibitor against HER1 (EGFR), HER2, and HER4.
* In vivo studies on HER2/3 expressing HCC PDX models suggest inhibition of pERB B2/3, pERK1 and pERK 2 with treatment with ASLAN001 (Varlitinib). Dose dependent inhibition of Cdc2 and pAKT in HCC PDX models treated with ASLAN001 (Varlitinib) also suggest robust inhibition of the PI3K pathway.
* EGFR overexpression in HCC and matched non tumor tissues were detected in (32.5%) and (28.6%), respectively. Moreover, missense and silent mutations were detected in (39.4%) and (33.3%) of HCC tissues, respectively.
* Determine the maximum tolerable dose (MTD) of ASLAN001 (Varlitinib) in advanced/metastatic HCC patients.
* After the recommended dose is determined, the Phase Ib portion of the study will evaluate the efficacy of ASLAN001 (Varlitinib) in HCC patients who have progressed on Sorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have unresectable or metastatic HCC with Childs Pugh status A with histologic confirmation.

   i) Subjects with only a radiologic diagnosis of HCC may be enrolled for screening in the study but histological confirmation is mandatory prior to the start of study therapy.

   ii) Evaluable tumor tissue (formalin-fixed, paraffin embedded archival or recent acquisition) must have 15 unstained slides for correlative studies. If archived samples are not available, subjects must consent to a pre-treatment fresh biopsy as a condition of protocol participation.
2. Patients must have failed Sorafenib or Lenvatinib due to disease progression or intolerance.
3. Presence of radiographically measurable disease based on RECIST v1.1.
4. No evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN).
5. Patients age ≥ 21 years at the time of written informed consent.
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Patient must be able to understand and willing to sign the informed consent form and donate tumor tissue (archival or fresh) for evaluation of relevant exploratory endpoints.
8. Patient with adequate organ and hematological function:

   a. Hematological function, as follows: i. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L ii. Platelet count ≥ 80 x 10^9/L b. Renal functions, as follows: i. Serum creatinine ≤ 1.5x ULN or eGFR > 60 mL/min/1.73m2 c. Hepatic function in addition to Childs Pugh score A: i. Total bilirubin ≤ 1.5 x ULN ii. AST and ALT ≤ 2.5 x ULN

Expansion cohort

1. Patients must agree to a post treatment biopsy
2. HER3 expression on IHC
3. Other inclusion criteria as above

Exclusion Criteria:

1. Patient with radiation or local treatment within the past 6 weeks for the target lesion(s).
2. Patients with major surgical procedures within 21 days prior to study entry.
3. Patient with brain lesion, known brain metastases (unless previously treated and well controlled for a period of at least 3 months).
4. Patient with malabsorption syndrome, diseases significantly affecting gastrointestinal function, resection of the stomach or small bowel, or difficulty in swallowing and retaining oral medications.
5. Patients with an uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, cardiac arrhythmia, diabetes, hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Patients with any history of other malignancy unless in remission for more than 1 year. (Non-melanoma skin carcinoma and carcinoma-in-site of uterine cervix treated with curative intent is not exclusionary).
7. Female patients who are pregnant or breast feeding.
8. Patients who were previously treated with ASLAN001 (Varlitinib).
9. Patients who have received any investigational drug (or have used an investigational device) within the last 14 days before receiving the first dose of study medication.
10. Patient with unresolved or unstable serious toxicity ( ≥ CTCAE 4.03 Grade 2) from prior administration of another investigational drug and/or prior cancer treatment.
11. Patients with a known history of HIV, decompensated cirrhosis, chronic active hepatitis or chronic persistent hepatitis.
12. Patients who need continuous treatment with proton pump inhibitors during the study period.
13. Any history or presence of clinically significant cardiovascular, respiratory, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease or any other condition which in the opinion of the Investigator could jeopardize the safety of the patient or the validity of the study results

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-05-05 (Estimated); Study Completion 2021-05-05 (Estimated)

PRIMARY OUTCOMES:
Definition of MTD (maximum tolerable dose) | up to 1 year since the start of treatment
  The maximum tolerable dose is defined as the highest evaluated dose where < 1/6 patients experiences DLT during the DLT evaluation window.

SECONDARY OUTCOMES:
Objective Response Rate | up to 1 year since the start of treatment
  Defined as the proportion of patients with a response of Partial Response or Complete Response, as defined by RECIST v1.1 criteria.
  Measurable disease:
  Tumor lesions: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of 10mm on CT scan Malignant lymph node: ≥15mm in short axis on CT scan Non-measurable disease: All other lesions, including small lesions (longest diameter <10mm or pathological lymph nodes with >10 to <15mm short axis) as well as truly non-measurable lesions
Progression Free Survival | up to 1 year since the start of treatment
  Defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression). Progression is defined in accordance with RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Raghav Sundar, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subbiah IM, Subbiah V, Tsimberidou AM, Naing A, Kaseb AO, Javle M, Fu S, Hong DS, Piha-Paul S, Wheler JJ, Hess KR, Janku F, Falchook GS, Wolff RA, Kurzrock R. Targeted therapy of advanced gallbladder cancer and cholangiocarcinoma with aggressive biology: eliciting early response signals from phase 1 trials. Oncotarget. 2013 Jan;4(1):156-65. doi: 10.18632/oncotarget.832. PMID 23391555
- [Background] Yang X, Wang W, Wang C, Wang L, Yang M, Qi M, Su H, Sun X, Liu Z, Zhang J, Qin X, Han B. Characterization of EGFR family gene aberrations in cholangiocarcinoma. Oncol Rep. 2014 Aug;32(2):700-8. doi: 10.3892/or.2014.3261. Epub 2014 Jun 13. PMID 24927194